CLINICAL TRIAL: NCT04542395
Title: Multilevel Participatory Intervention to Reduce Barriers and Promote Social and Behavioral Facilitators of COVID-19 Testing Among African Americans and Latinx Public Housing Residents
Brief Title: COVID-2019 Testing and Vaccination Among African American and Latinx Public Housing Residents
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not funded
Sponsor: Charles Drew University of Medicine and Science (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: COVID19testingvacc
Record Dates: First submitted 2020-09-03; First posted 2020-09-09 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Coronavirus
MeSH Terms: conditions — Coronavirus Infections | interventions — Vaccination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Increasing Uptake of COVID-19 Testing and Vaccination (Experimental): This is a pre-experimental "one group pretest-posttest" design to improve COVID-19 associated health outcomes and willingness and uptake toward testing and vaccination among 310 Hispanic and African American public housing residents in South Los Angeles. The proposed intervention will employ (1) culturally sensitive, (2) theoretically based intervention that will be jointly delivered by our COVID-19 health ambassadors and our researchers. We will use the Information, Motivation, and Behavioral Skills (IMB) model and the Transtheoretical Model to implement the intervention.
  Interventions: Behavioral: Increasing Willingness and Uptake of COVID-19 Testing and Vaccination

INTERVENTIONS:
Behavioral: Increasing Willingness and Uptake of COVID-19 Testing and Vaccination — Provide/enhance knowledge, modify attitudes, motivate and provide skills and resources to reduce COVID-19 related risk and challenges and increase willingness and uptake in COVID-19 testing and vaccination.

SUMMARY:
This proposal seeks to enhance acceptability and uptake of COVID-19 testing and vaccination to engage African American and Latinx public housing residents in South Los Angeles. Given the multiple disparities experienced by public housing residents, the investigators will utilize a theoretically-based, multidisciplinary and culturally tailored intervention to reduce barriers and implement innovate strategies to engage this population in the uptake of COVID-19 testing and vaccination.

DETAILED DESCRIPTION:
Through the engagement and empowerment of 15 trained COVID-19 health ambassadors, the investigators will jointly implement and evaluate a theoretically based and culturally-sensitive socio-behavioral intervention that will: a) reduce mistrust, fatalistic beliefs, and related psychosocial barriers that hinder COVID-19 testing and vaccination; b) increase receptivity and willingness for uptake of COVID-19 testing and vaccination; and c) assess perceived impact of psychosocial and health outcomes related to COVID-19 testing and vaccination for 310 African American and Latinx public housing residents.

ELIGIBILITY:
Inclusion Criteria:

* Identify as Latino/Hispanic or African American/Black
* Reside in one of the six collaborating public housing
* 18 years old and older
* Speak either English or Spanish

Exclusion Criteria:

* Does not self-identify as African American and/or Black
* Under the age of 18
* Unable to speak English or Spanish
* Does not Reside in one of the six collaborating public housing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of COVID-19 testing, pneumococcal and influenza vaccinations Using Test History Self-Report | Intervention: 3 months; Follow-up Point: 6 months post-intervention
  By comparison of pre-, post- intervention, and six-months follow-up data, we anticipate the following compared to baseline: a 30% change in willingness and uptake for testing and vaccination.
Percentage of Participants Achieving Decreased Levels of COVID-19 Risk Using the NIH Toolbox Surveys on COVID-19 | Intervention: 3 months; Follow-up Point: 6 months post-intervention
  By comparison of pre-, post- intervention, and six-months follow-up data, we anticipate the following compared to baseline: a 30% change in perceived COVID-19 risk.
Percentage of Participants Achieving Decreased Levels of COVID-19 Mistrust and Barriers Using the NIH Toolbox Surveys on COVID-19 | Intervention: 3 months; Follow-up Point: 6 months post-intervention
  By comparison of pre-, post- intervention, and six-months follow-up data, we anticipate the following compared to baseline: a 40% change in mistrust and perceived barriers toward COVID-19 testing and vaccination,

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen Bazargan, PhD, Principal Investigator — Charles R. Drew University of Medicine & Science
Locations (1):
- Housing Authority of Clty of Los Angeles, Los Angeles, California, United States